CLINICAL TRIAL: NCT04434183
Title: Comparison of the Effects of Home Exercise Program and Isokinetic Exercise Program on Pain, Muscle Strength, Functionality, Sense of Proprioception and Quality of Life in Subacromial Impingement Syndrome Patients
Brief Title: Comparison of the Effects of Home Exercise and Isokinetic Exercise Program in Subacromial Impingement Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Sevgi Atar, Administrative Director of PMR Clinic, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 851
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Home Exercise; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- isokinetic exercise (Active Comparator): The group (isokinetic exercise group, n = 25) was given isokinetic exercise.
  Interventions: Device: Exercises of rehabilitation
- home exercise (Active Comparator): The group(home exercise group, n=25) was given home exercise program.
  Interventions: Device: Exercises of rehabilitation

INTERVENTIONS:
Device: Exercises of rehabilitation — Compare and evaluate of the effects of the routin physical medicine and rehabilitation programs in impingement patients
  Other Names: Isokinetic cybex dynamometer

SUMMARY:
The aim of this study is to evaluate and compare the effects of home exercise program and isokinetic exercise program on pain, muscle strength, functionality, proprioception sensation and quality of life in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
The study was designed prospectively. A total of 50 patients with subacromial impingement syndrome according to clinical and MRI findings with shoulder pain for at least 3 months were included in the study. Patients were randomly divided into two groups. The first group (isokinetic exercise group, n = 25) was given isokinetic exercise. The second group(home exercise group, n=25) was given home exercise program. Patients were evaluated before and after treatment and 3 months after the end of treatment. In the evaluation, VAS, Shoulder Pain and Disability Index, Constant Murley Scoring, Shoulder Disability Questionnaire, Health Assessment Questionnaire, Pittsburgh Sleep Quality Index, Humic Norm II isokinetic device were used. At statistically evaluation of data Student T Test and Mann Whitney U tests were used. In qualitative datas comparison Ki-Kare Test was used. Significance was evaluated at the level of p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain and functional disability at least 6 months

Exclusion Criteria:

* Instability of shoulder, Stage 2-3 adhesive capsulitis, tendinitis or bursitis, cervical radiculopathy, underwent surgery, norological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Assessment of shoulder examination findings | 3 months
  The investigators evaluated to pre-treatment, intermediate post-treatment, and late post-treatment shoulder examination findings. The investigators used to painful arc test consisting of 13 questions that scored from zero to ten.
Assessment of shoulder functions | 3 months
  The investigators evaluated to pre-treatment, intermediate post-treatment, and late post-treatment shoulder functions and muscle strenght. The investigators used to Constant-Murley functional evaluate scale consisting of four parameters that scored from zero to one hundered.
Assessment of muscle strenght | 3 months
  The investigators evaluated it with isokinetic cybex dynamometer. The isokinetic cybex dynamometer assessments using newton-meter for muscle strenght and angle degree for velocity measurements.
Assessment of quality of life | 3 months
  The investigators evaluated to pre-treatment, intermediate post-treatment, and late post-treatment quality of life values with Pittsburg sleep quality index. The Pittsburg sleep quality index consisting of 23 questions that scored from zero to three.
Assessment of sense of proprioseption | 3 months
  The investigators evaluated it with isokinetic cybex dynamometer. The isokinetic cybex dynamometer assessments using angle degree for sense of position.
Assessment of shoulder pain | 3 months
  The investigators evaluated to pre-treatment, intermediate post-treatment, and late post-treatment for shoulder pain. The investigators used to visual analog score for pain that scored from zero to ten.
Assessment of shoulder disability | 3 months
  The investigators evaluated to pre-treatment, intermediate post-treatment, and late post-treatment for shoulder disability. The investigators used to shoulder disability questionnare consisting of 16 questions that scored yes or no. Calculation; score = [Yes counts / (Yes counts + No counts)]x100. The score seems, zero point is maximal fine health and 100 points (maximal point) is poor health.
Assessment of physical health situation | 3 months
  The investigators evaluated to pre-treatment, intermediate post-treatment, and late post-treatment for physical health situation. The investigators used to health evaluated inventory. The inventroy consisting of 20 questions that scored from zero to three per question. Zero point is maximal fine health and 60 points are maximal poor health.

CONTACTS AND LOCATIONS:
Overall Officials: OMER KURU, FULL PROF, Study Chair — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akman S, Kucukkaya M. [Subacromial impingement syndrome: pathogenesis, clinical features, and examination methods]. Acta Orthop Traumatol Turc. 2003;37 Suppl 1:27-34. Turkish. PMID 14578662
- [Result] Campbell RS, Dunn A. External impingement of the shoulder. Semin Musculoskelet Radiol. 2008 Jun;12(2):107-26. doi: 10.1055/s-2008-1078699. PMID 18509791
- See also: Subacromial Impingement Syndrome: Pathogenesis, Clinical Features, and Examination Methods — https://pubmed.ncbi.nlm.nih.gov/14578662/
- See also: External Impingement of the Shoulder — https://pubmed.ncbi.nlm.nih.gov/18509791/?from_single_result=Campbell+RS%2C+Dunn+A%3A+External+impingement+of+the+shoulder.